



IRAS ID: 242462

## **Informed Consent Form**

## Assessing gut permeability using spectroscopy

Study title: Non-invasive transcutaneous spectroscopy for the assessment of gut permeability (GutPerm)

IRAS Project ID: 242462

| Pa | atient Trial ID Number: | |
|---|---|---|
| Na | ame of Principal Investigator: <u>Dr Alex Thompson</u> | |
| Na | ame of patient to whom this ICF applies: | |
| | Please | initial boxes |
| 1. | I confirm that I have read and understand the Patient Information Sheet "Assessing gut permeability using spectroscopy v4.2A 01-May-2019" for the above study and have had the opportunity to ask questions about the study and understand what is involved. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or other legal rights being affected, and I understand that any remaining samples will be destroyed at my request, but data collected up to the point of my withdrawal may still be used. | |
| 3. | If I have had an intestinal biopsy as part of my routine clinical care, I am happy for some of my tissue, if surplus to clinical need, to be given to the research team and/or approved collaborators within and outside the European Economic Area for healthcare and/or medical research purposes. I am also happy for any clinical data obtained from these biopsies and samples to be accessed and used by the research team. | |
| 4. | I agree to have a 'Spectroscopic gut permeability test' and understand that there is a small risk of nausea and other allergic reactions (including anaphylaxis) with this test. | |
| 5. | I agree to provide two 5 ml blood samples during my study visit (equivalent to approximately one teaspoon of blood for each sample). | |
| | If you do <u>NOT</u> consent to provide two 5 ml blood samples, please put a line through all of point 5 above, and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | |
| 6. | I agree to provide two urine samples during my study visit. | |
| | If you do <u>NOT</u> consent to provide two urine samples, please put a line through all of point 6 above, and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | |
| 7. | I agree to provide one or more stool samples within approximately 48 hours of my study visit. | |
| | If you do $\underline{NOT}$ consent to collection of stool samples, please put a line through all of point 7 above, and do $\underline{NOT}$ initial the box as indicated – you can still participate in the main trial. | |
| 8. | I agree to have a 'PEG permeability test' and understand that there is a small risk of diarrhoea and bloating with this test. | |

## Imperial College London



| 9. | from Imperial College Healthcare I | NHS Trust, from Impe<br>my taking part in this | ay be looked at by authorised individuals<br>rial College London, or from regulatory<br>s research. I give permission for these | , |
|---|---|---|---|---|
| 10. | | outside the European | alysed, reported and transferred to other<br>n Economic Area for healthcare and/or<br>will remain anonymous. | |
| 11. | of this study to be used in future re<br>approval from an independent resea | esearch projects that our<br>arch ethics committee.<br>Area. Under these circ | samples that I give that are used as part<br>comply with regulations and which have<br>This may include transfer of my samples<br>cumstances my samples will be retained<br>egulated Biobank. | |
| | | | nd used for future research in this way,<br><u>OT</u> initial the box as indicated – you can | |
| 12. | 2. I give consent for the research team to inform my general practitioner (GP) of my participation in the study. | | | |
| 13. | 3. I wish to be contacted by e-mail with a summary of the research findings once the study is complete. Your e-mail address will not be used for any other purpose. | | | |
| | Contact e-mail: | | | |
| | If you do <u>NOT</u> wish to be contacted regarding the study results, please put a line through all of point 13 above, do <u>NOT</u> leave a contact e-mail address and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | | | |
| 14. | 14. I agree to take part in the study. | | | |
| Ple | ase sign and date below. | | | |
| Nar | me of Subject | Signature | Date | |
| <br>Nar | me of Person taking consent | Signature | <br>Date | |

1 copy for subject; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes

IRAS ID: 242462